CLINICAL TRIAL: NCT01389128
Title: Application of Non-pharmacological Resources in Assisting Labor: Randomized Controlled Trial
Brief Title: Non-pharmacological Resources in Assisting Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvana Maria Quintana, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FR443033
Record Dates: First submitted 2011-06-30; First posted 2011-07-07 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Labour Pain
Keywords: labor; pain; massage; natural birth
MeSH Terms: conditions — Labor Pain; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Pregnant women who receive assistance from the routine CRSM MATER care, not being assisted by the physiotherapist, but that will be evaluated at the same time in the intervention group.
  Interventions: Other: Routine care
- Intervention Group (Experimental): Pregnant women who receive the application the combination of non-pharmacological resources according to cervical dilation: pelvic mobility , lumbosacral massage and warm shower.
  Interventions: Other: Non-pharmacological resources

INTERVENTIONS:
Other: Non-pharmacological resources — A sequence of non-pharmacological resources were applied to the patient by the researcher according to uterine cervical dilation, as follows:
  * Pelvic mobility on the exercise ball oriented and accompanied by the researcher for 40 minutes;
  * Lumbosacral massage for a period of 40 minutes, when dilation was between 5 and 6 cm. During the procedure, the woman in labor was allowed to freely choose the most comfortable position; and,
  * Warm shower with the water flow directed to the lower-back of the woman in labor, for 40 minutes, when uterine cervical dilation was equal to or higher than 7cm.
  Arms: Intervention Group
Other: Routine care — Routine care of the institution performed by the staff, without the presence of the researcher that included offering a balanced meal, continuous support with the presence of a partner or family throughout labor, use of oxytocin when prescribed by the staff, use of drug analgesia when requested by the patient.
  Arms: Control Group

SUMMARY:
The proposed project will be conducted to evaluate the influence of application resources associated with non-pharmacological during labor for pain relief and accelerated phase of expansion. Although mothers' access to resources for non-pharmacological pain relief during labor is recommended, is not seen as the application of routine obstetric practice, although it has been demonstrated benefits and scientific evidence with your application. It is believed that the implementation of associated application of non-pharmacological resources in assisting the labor can be introduced into daily practice in various hospitals in the country, minimizing pain and favoring the shorter duration of labor, decrease in use of painkillers and inductors, resulting in a reduction of complications, improves the comfort of the mother making her birth experience more satisfying and rewarding, being assisted with security and trained by multidisciplinary teams.

DETAILED DESCRIPTION:
The current model of care delivery has demanded a technical-assistance approach that prioritizes the quality of care, as indissolubly concerns the employment of technology, knowledge, the centrality of dialogue between professionals and patients and individualized choice resources deemed suitable for safe delivery. Seeking to implement a less interventionist care with evidence-based practice and greater incentive to vaginal delivery, the programs were created humanization of labor and birth, with the use of various non-pharmacological resources. This study aimed to evaluate the effectiveness of the combination of non-pharmacological resources during the dilation in relieving the pain of the mothers. The research will be of type randomized controlled trial, consisting of low-risk primigravidae admitted at the Reference Center for Women's Health in Ribeirão Preto. The mothers will be distributed in two groups (intervention protocol features non-drug) and Control (routine maternity) and will be evaluated before and after application of each resource, and the control group in the same time according to cervical dilation. Evaluation will be conducted by a visual analog scale and / or facial pain and pain location diagram and postpartum will be applied a validated questionnaire Experience and Satisfaction with childbirth. After collecting the data, the groups are statistically analyzed using the linear regression model with mixed effects (fixed and random), taking into account a value of p <0.05 to obtain the statistical significance of 5%.

ELIGIBILITY:
Inclusion Criteria:- Agreed to participate in the study after reading and signing the consent form;

* Primigravida;
* Pregnancy only;
* Gestational age ≥ 37 weeks;
* Presentation fetal head
* Chorioamniotic intact membranes
* Working with spontaneous onset of labor
* Admission at the beginning of active phase dilation (4-5 cm)
* Lack of maternal and fetal pathologies
* Literacy - primary education
* Absence of cognitive problems

Exclusion Criteria:

* Pregnant women admitted for induction of labor
* Rupture premature or early of chorioamniotic membranes
* Use of uterotonic drugs before the active phase

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvana M Quintana, professor, Principal Investigator — Faculty of Medicine of São Paulo University
Locations (1):
- Referral Center Women's Health - Mater, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Huntley AL, Coon JT, Ernst E. Complementary and alternative medicine for labor pain: a systematic review. Am J Obstet Gynecol. 2004 Jul;191(1):36-44. doi: 10.1016/j.ajog.2003.12.008. PMID 15295342
- [Derived] Gallo RBS, Santana LS, Marcolin AC, Duarte G, Quintana SM. Sequential application of non-pharmacological interventions reduces the severity of labour pain, delays use of pharmacological analgesia, and improves some obstetric outcomes: a randomised trial. J Physiother. 2018 Jan;64(1):33-40. doi: 10.1016/j.jphys.2017.11.014. Epub 2017 Dec 27. PMID 29289579

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control Group (CG): Pregnant women who receive assistance from the routine CRSM MATER care, not being assisted by the physiotherapist, but that will be evaluated at the same time in the intervention group.
  Control Group: Routine care of the institution performed by the staff, without the presence of the researcher
- Intervention Group: Intervention Group (IG): Pregnant women who receive the application the combination of non-pharmacological resources: standing upright pelvic mobility in the ball (4 to 5 cm), alternating stance associated with lumbosacral massage (5 and 6 cm) and shower (>or= 7 cm);
  Intervention Group: application of the combination of non-pharmacological resources: standing upright pelvic mobility in the ball, alternating stance associated with lumbosacral massage and shower;
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 40 | 40
Completed | 35 | 34
Not Completed | 5 | 6
Not completed — Fetal distress | 1 | 0
Not completed — Cervix dilation stop | 1 | 2
Not completed — Rapid labor evolution | 3 | 2
Not completed — Intolerance to procedure | 0 | 2

BASELINE CHARACTERISTICS:
Population: Low-risk primigravidae women admitted to the maternity ward in the active phase of labor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.85 (4.22) | 20.60 (4.14) | 20.72 (4.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kilograms per square meter] | 28.4 (5.36) | 26.9 (3.72) | 27.65 (4.54)
School degree [Count of Participants; unit: Participants]
  Elementary School | 13 | 11 | 24
  High School | 24 | 25 | 49
  College degree | 3 | 4 | 7
Marital status [Count of Participants; unit: Participants]
  single | 6 | 3 | 9
  married | 11 | 14 | 25
  stable union | 23 | 23 | 46
Preparation for labour [Number; unit: participants]
  yes | 10 | 11 | 21
  no | 30 | 29 | 59
Presence of partner [Count of Participants; unit: Participants] — The measure refers to the number of participants who were accompanied by a partner or family member throughout labor
  Participants | 40 | 40 | 80
Occupation [Count of Participants; unit: Participants]
  unemployed | 23 | 29 | 52
  employed | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief
Description: The Visual Analogue Scale - VAS - was used to measure the intensity of the pain described by the patients during the study. The patient was requested do mark a dot in a straight line, measuring 100mm, being a 0 (Zero) no pain and 100 the most intense pain. The researcher then would measure the estimated pain intensity in millimeters. The pain intensity was measured in all three phases before and after each procedure assigned to each group. The phases and their respective procedures were:
  * Phase I: 4-5cm of cervical dilation (pelvic mobility in exercise ball)
  * Phase II: 5-6cm of cervical dilation (lumbosacral massage)
  * Phase III: 7cm or higher cervical dilation (warm shower)
Time Frame: ten hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
millimeters
  Phase I - Before | 79.5 (18.1) | 73.8 (16.2)
  Phase I - After | 71.0 (35.0) | 51.7 (19.5)
  Phase II - Before | 75.6 (40.8) | 83.6 (15.8)
  Phase II - After | 36.3 (39.7) | 67.3 (24.3)
  Phase III - Before | 75.9 (37.0) | 96.4 (8.5)
  Phase III - After | 54.1 (34.2) | 60.6 (25.5)

2. Secondary Outcome: Evolution of Labor
Description: Amount of minutes, from admission to labor.
Time Frame: 10 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Control Group: Routine care of the institution
- Intervention Group: Combined and sequential non-pharmacological resources
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
minutes | 492 (35) | 382 (24)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Other; p < 0.01, Chi-squared

3. Secondary Outcome: Moment That Women Requested Analgesia During the Active Phase of Labor
Description: Mean uterine cervical dilation at the moment the patient requested analgesia for pain relief. Data obtained from medical record
Time Frame: 10 hours
Measure: Mean (Standard Deviation); unit: centimeter
Groups:
- Control Group: Control Group: Routine care of the institution performed by the staff, without the presence of the researcher
- Intervention Group: Intervention Group: application of the combination of non-pharmacological resources: standing upright pelvic mobility in the ball, alternating stance associated with lumbosacral massage and shower;
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
centimeter | 6 (1) | 8 (0.8)

4. Secondary Outcome: Number of Women Who Received Pharmacological Analgesia
Description: Determine the number of women who where submitted to pharmacological analgesia, either prescribed by the attending physician ou requested by the patient herself.
Time Frame: 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 37 | 34

5. Secondary Outcome: Type of Delivery
Description: Type of delivery at the end of the active phase of labor.
Time Frame: 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  Vaginal | 30 | 35
  C-Section | 10 | 5
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Other; p = 0.68, Chi-squared

6. Secondary Outcome: Number of Participants Whose Neonates Had:
Description: Number and type of neonatal complications as reported in medical chart
Time Frame: 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  Shoulder dystocia | 1 | 0
  Fetal respiratory distress | 6 | 0
  No complications | 33 | 40

7. Secondary Outcome: Number of Participants With:
Description: Number and type of maternal complications as reported in medical chart
Time Frame: 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants
  Rapid evolution of labor | 3 | 2
  Hypotension | 1 | 0
  Dilation stop | 6 | 3
  Fetal descent stop | 3 | 1
  Intrapartum hemorhage | 0 | 1
  No complications | 27 | 33

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 7/40 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Intervention Group (N=40)
Neonate complications (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 0 (0) — When neonates suffered shoulder dystocia or respiratory distress

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No